CLINICAL TRIAL: NCT05317936
Title: Pirtobrutinib (LOXO-305) Consolidation for MRD Eradication in Patients With Chronic Lymphocytic Leukemia/Small Lymphocytic Lymphoma (CLL) Treated With Venetoclax
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: <75% participation
Sponsor: M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2021-0953; NCI-2022-02427 (Other: NCI-CTRP-Clinical Trial Reporting Registry)
Record Dates: First submitted 2022-03-15; First posted 2022-04-08 (Actual); Last update posted 2025-12-15 (Actual); Status verified 2025-12

CONDITIONS: Chronic Lymphocytic Leukemia; Small Lymphocytic Lymphoma
MeSH Terms: conditions — Leukemia, Lymphocytic, Chronic, B-Cell | interventions — pirtobrutinib; venetoclax

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Pirtobrutinib+venetoclax (Experimental): Pirtobrutinib by mouth at the same time each day Venetoclax by mouth at the same time each day.
  Interventions: Drug: Pirtobrutinib; Drug: Venetoclax

INTERVENTIONS:
Drug: Pirtobrutinib — Given by PO
  Other Names: LOXO-305
Drug: Venetoclax — GIven by PO
  Other Names: ABT-199; GDC-0199

SUMMARY:
To learn if the combination of LOXO-305 (pirtobrutinib) and venetoclax can help to control previously treated chronic lymphocytic leukemia/small lymphocytic lymphoma (CLL/SLL).

DETAILED DESCRIPTION:
Primary Objective:

I. To estimate the therapeutic efficacy of pirtobrutinib consolidation in patients who have detectable CLL in peripheral blood after receiving venetoclax for at least 12 cycles. The primary endpoint will be the rate of undetectable MRD (U-MRD4) in the peripheral blood, assessed by NGS at a threshold of 0.01% sensitivity, after 24 cycles of combination therapy.

SECONDARY OBJECTIVES:

I. Determine the complete remission (CR)/complete remission with incomplete marrow recovery (CRi) rate after 6, 12 18 and 24 cycles of combination therapy, in patients who were not in CR/CRi at study initiation and estimate the time to best response with this combination.

II. Determine the cumulative rate of blood and bone marrow minimal residual disease undetectable minimal residual disease (MRD) by next generation sequencing (NGS) at thresholds of 0.01% sensitivity (MRD4), 0.001% sensitivity (MRD5) and 0.0001% sensitivity (MRD6).

III. Achievement of undetectable MRD at a sensitivity of 0.0001% (MRD6) in the bone marrow in patients who achieve undetectable (U)-MRD6 in peripheral blood.

IV. Determine the safety of combined pirtobrutinib and venetoclax. V. Determine the progression-free and overall survival.

OUTLINE:

Patients receive pirtobrutinib orally (PO) once daily (QD) and venetoclax PO QD on days 1-28. Treatment repeats every 28 days for up to 24 cycles in the absence of disease progression or unacceptable toxicity. After 24 cycles of combination therapy, patients who achieve U-MRD4 discontinue therapy. Patients who do not achieve U-MRD4 receive pirtobrutinib PO QD on days 1-28. Treatment repeats every 28 days for up to 36 cycles in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up at 4 weeks, and then every 24 weeks (6 months) for up to 5 years.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of CLL per International Workshop on Chronic Lymphocytic Leukemia (IWCLL) 2018 criteria
* Received venetoclax for at least 12 cycles, with MRD > 0.01% detectable in peripheral blood, by Adaptive Biotechnologies NGS assay, within the month prior to study enrollment
* Age 18 years or older
* Eastern Cooperative Oncology Group (ECOG) performance status =< 2
* Serum bilirubin =< 1.5 x upper limit of normal (ULN) or =< 3 x ULN for patients with Gilbert's disease
* Serum creatinine clearance of >= 30 ml/min (calculated or measured)
* Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) =< 3.0 x ULN, unless clearly due to documented disease involvement, in which case ALT and AST =< 5.0 x ULN
* Platelet count of >= 50,000/ul, with no platelet transfusion in prior 2 weeks
* Absolute neutrophil count (ANC) >= 1000/ul in the absence of growth factor support
* Hemoglobin >= 8 mg/dL
* Activated partial thromboplastin time (aPTT) or partial thromboplastin time and prothrombin time (PT) or international normalized ratio (INR) not greater than 1.5 x ULN
* Ability to provide informed consent and adhere to the required follow-up
* Women of childbearing potential must have a negative serum or urine beta human chorionic gonadotropin (beta-hCG) pregnancy test result within 7 days prior to the first dose of study drugs and must agree to use use both a highly effective method of birth control (e.g., implants, injectables, combined oral contraceptives, some intrauterine devices [IUDs], complete abstinence, or sterilized partner) and a barrier method (e.g., condoms, vaginal ring, sponge, etc) during the period of therapy and for 6 months after the last dose of study drug. Women of non-childbearing potential are those who are postmenopausal (defined as absence of menses for >= 1 year) or who have had a bilateral tubal ligation or hysterectomy. Men who have partners of childbearing potential must agree to use effective contraception, defined above, during the study and for 30 days following the last dose of study drug

Exclusion criteria Exclusion Criteria:

* Known or suspected Richter's transformation to diffuse large B cell lymphoma (DLBCL), prolymphocytic leukemia, or Hodgkin lymphoma at any time preceding enrollment
* Known or suspected history of central nervous system (CNS) involvement by CLL
* History of grade >= 3 arrhythmia on prior covalent Bruton's tyrosine kinase (BTK) inhibitor
* Patients who experienced a major bleeding event on a prior BTK inhibitor

  * NOTE: Major bleeding is defined as bleeding having one or more of the following features: life-threatening bleeding with signs or symptoms of hemodynamic compromise; bleeding associated with a decrease in the hemoglobin level of at least 2 g/dL; or bleeding in a critical area or organ (e.g., retroperitoneal, intraarticular, pericardial, epidural, or intracranial bleeding or intramuscular bleeding with compartment syndrome)
* Active second malignancy. Patients with a treated second malignancy and with likelihood of requiring systemic therapy within the next 2 years of < 10%, as determined by an expert in the field, will be eligible. Examples include:

  * Adequately treated non-melanomatous skin cancer or lentigo maligna melanoma without current evidence of disease
  * Adequately treated cervical carcinoma in situ without current evidence of disease
  * Localized (e.g., lymph node negative) breast cancer treated with curative intent with no evidence of active disease present for more than 3 years and receiving adjuvant hormonal therapy
  * Localized prostate cancer undergoing active surveillance
  * History of treated and cured Hodgkin's disease or non-Hodgkin lymphoma (NHL) < 5 years from diagnosis
* Major surgery within 4 weeks of planned start of study therapy
* A significant history of renal, neurologic, psychiatric, endocrine, metabolic or immunologic disorder, that, in the opinion of the Investigator, would adversely affect the patient's participation in this study or interpretation of study outcomes
* History of allogeneic or autologous stem cell transplant (SCT) or chimeric antigen receptor (CAR)-T therapy within the past 60 days or presence of any of the following, regardless of prior SCT and/or CAR-T therapy timing:

  * Active graft versus host disease (GVHD)
  * Need for anti-cytokine therapy for toxicity from CAR-T therapy
  * Residual symptoms of neurotoxicity > grade 1 from CAR-T therapy
* Active uncontrolled auto-immune cytopenia (e.g., autoimmune hemolytic anemia [AIHA], idiopathic thrombocytopenic purpura [ITP])
* Significant cardiovascular disease, defined as any of the following:

  * Unstable angina or acute coronary syndrome within the past 2 months
  * History of myocardial infarction within 6 months prior to planned start of study treatment
  * Documented left ventricular ejection fraction (LVEF) by any method of =< 45% in the 12 months prior to planned start of study treatment
  * >= grade 3 New York Heart Association (NYHA) functional classification system of heart failure
  * Uncontrolled or symptomatic arrhythmias
* Prolongation of the QT interval corrected (QTc) for heart rate using Fredericia's Formula (QTcF) > 470 msec on an electrocardiogram (EKG) during screening

  * QTcF is calculated using Fredericia's Formula
  * Correction of suspected drug-induced QTcF prolongation or prolongation due to electrolyte abnormalities can be attempted at the Investigator's discretion, and only if clinically safe to do so with either discontinuation of the offending drug or switch to another drug not known to be associated with QTcF prolongation or electrolyte supplementation
  * Correction of QTc for underlying bundle branch block (BBB) permissible
* Hepatitis B or hepatitis C testing indicating active/ongoing infection based on screening laboratory tests as defined as:

  * Hepatitis B virus (HBV): Patients with positive hepatitis B surface antigen (HBsAg) are excluded. Patients with positive hepatitis B core antibody (anti-HBc) and negative HBsAg require hepatitis B polymerase chain reaction (PCR) evaluation. Patients who are hepatitis B PCR positive will be excluded
  * Hepatitis C virus (HCV): positive hepatitis C antibody. If positive hepatitis C antibody result, patient will need to have a negative result for hepatitis C ribonucleic acid (RNA) before randomization. Patients who are hepatitis C RNA positive will be excluded
* Evidence of other clinically significant uncontrolled condition(s) including, but not limited to, uncontrolled systemic infection (viral, bacterial, or fungal) or other clinically significant active disease process which in the opinion of the Principal Investigator may pose a risk for patient participation. Screening for chronic conditions is not required
* Known human immunodeficiency virus (HIV) infection, regardless of CD4 count. Patients with unknown or negative status are eligible
* Known active cytomegalovirus (CMV) infection. Patients with unknown or negative status are eligible
* Clinically significant active malabsorption syndrome or other condition likely to affect gastrointestinal (GI) absorption of the oral administered study treatments
* Investigational agent or anti-cancer therapy other than venetoclax, with the exception of hormonal therapy for breast or prostate cancer. Other agents must be discontinued for at least 4 weeks for monoclonal antibody therapy or 5 half lives for other agents
* Use of > 20 mg prednisone QD or equivalent dose of steroid per day at the time of cycle 1 day 1 (C1D1). Patients may not be on prednisone of any dose intended for anti-neoplastic use
* Patients requiring therapeutic anticoagulation with warfarin or another Vitamin K antagonist
* Current treatment with strong cytochrome P450 (CYP) 3A4 (CYP3A4) inducers and/or strong P-glycoprotein (P-gp) inhibitors. Because of their effect on CYP3A4, use of any of the following within 3 days of study treatment start or planned use during study participation is prohibited:

  * Grapefruit or products from grapefruit
  * Seville oranges or products from Seville oranges
  * Star fruit or products from star fruit
* Vaccination with a live vaccine within 28 days prior to study start
* Previous treatment with another non-covalent BTK inhibitor, such as nemtabrutinib
* Pregnancy, lactation or plan to breastfeed during the study or within 30 days of the last dose of study treatment
* Patients with known hypersensitivity to any component or excipient of LOXO-305 and venetoclax
* Any unresolved toxicity from prior therapy greater than Common Terminology Criteria for Adverse Events (CTCAE) (version 5.0) grade 2 at the time of starting study treatment, except for alopecia

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2022-11-16 (Actual); Primary Completion 2025-10-06 (Actual); Study Completion 2025-10-06 (Actual)

PRIMARY OUTCOMES:
Rate of undetectable (U) minimal residual disease (MRD) in the peripheral blood | Up to completion of cycle 24 (each cycle is 28 days)
  Assessed by next generation sequencing (NGS) at a threshold of 0.01% sensitivity. The rate of U-MRD will be reported separately for each cohort, along with the corresponding exact 95% confidence interval.

CONTACTS AND LOCATIONS:
Overall Officials: Alessandra Ferrajoli, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- M D Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: M D Anderson Cancer Center — http://www.mdanderson.org

DOCUMENTS (1):
  • Informed Consent Form (2023-05-26): https://cdn.clinicaltrials.gov/large-docs/36/NCT05317936/ICF_000.pdf